CLINICAL TRIAL: NCT06621992
Title: Skills to Enhance Positivity in Young Adults
Acronym: STEP YA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 016816
Record Dates: First submitted 2024-09-30; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Positive Affect; Mindfulness; Gratitude; Savoring; Depression
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skills to Enhance Positivity (Experimental): Participants received 4 group sessions, session 1 focused on positive affect psychoeducation, session 2 on mindfulness, 3 on savoring and 4 on gratitude. Once completing the group sessions participants received text messages for 1 month before tapering off.
  Interventions: Other: Skills to Enhance Positivity
- Treatment as Usual (Active Comparator): Participants received their standard treatment as usual
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Other: Skills to Enhance Positivity
  Arms: Skills to Enhance Positivity
Other: Treatment as Usual — Participants received treatment as usual
  Arms: Treatment as Usual

SUMMARY:
The goal of this study is to test the feasibility and acceptability of a positive affect intervention for suicide in a population of young adults. Skills to Enhance Positivity (STEP) has been demonstrated to be feasible and acceptable among adolescents when delivered individually. The current study aims to test feasibility and acceptability in a group setting of young adults. The specific aims of STEP also seek to establish whether participants who received STEP report a significant increase in attention towards positive affect compared to those receiving Treatment As Usual (TAU). They also seek to explore whether participants who received STEP will report a significant decrease in suicidal ideation and depression compared to those receiving TAU. The final aim is to explore whether an increase in attention to positive affect regardless of condition is a potential mechanism of change for reductions in suicidal ideation and depression. Participants will be randomized into STEP or TAU groups, they will complete baseline and follow-up assessments after a period of 3-months. Participants enrolled in STEP will receive in-person group sessions focusing on psychoeducation of positive affect as well as skills in mindfulness, gratitude and savoring designed to promote positive affect. After completing the group sessions they will also receive text messages for one month, where they will receive prompts to practice skills they learned in the group setting.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a recent history of depression and are English-speaking
* Participants also must have a cell phone with text-messaging capabilities

Exclusion Criteria:

* Participants who have acute psychotic disorders or cognitive deficits that would preclude full understanding of the protocol, intervention and assessment materials

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Feasibility and Acceptability of a group intervention | Will be assessed at follow-up at 3-months
  Feasibility and acceptability will be evaluated using self-report questionnaires and interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request to Principal Investigator
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon request
Access Criteria: Upon request